CLINICAL TRIAL: NCT00405743
Title: A Phase I/II Study of CP-4055 in Patients With Refractory/Relapsed Hematologic Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clavis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP4055-106
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Hematologic Malignancies; AML
Keywords: CP-4055; ELACYT™; Cancer; Refractory; Relapsed; Hematologic Malignancies; Leukemia; ALL; AML; AMM; CLL; CML; CMML; MDS
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms; Recurrence; Leukemia | interventions — 5'-oleoyl cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): CP4055, 2 and 4 hour IV infusion
  Interventions: Drug: CP-4055
- Arm B (Experimental): CP-4055, Continuous IV infusion
  Interventions: Drug: CP-4055

INTERVENTIONS:
Drug: CP-4055 — CP-4055 Continuous IV infusion
  Arms: Arm B
Drug: CP-4055 — CP4055 2 and 4 hour IV infusion
  Arms: Arm A

SUMMARY:
Patients with refractory or relapsed hematologic malignancies will receive CP-4055 intravenously(IV) on Day 1-5 every three weeks until complete response or disease worsening/progressing

DETAILED DESCRIPTION:
This is a multicentre clinical study conducted in the USA and in Europe. It is an open label, dose escalation study designed to characterize the safety, tolerability, pharmacokinetics (PK), and efficacy of CP-4055 as a single agent when administered as a 2 hours intravenous (IV) or a continuous IV (CIV) infusion administered daily for 5 days in a 21-day cycle, either alone or with idarubicin IV, in patients with refractory/relapsed hematologic malignancies who have either failed potentially curative therapy or are considered unsuitable for standard therapy.

In a second phase of the study the efficacy of single agent CP-4055 in patients with AML may be assessed.

It is intended that patients receive a minimum of two cycles of therapy in the absence of unacceptable toxicity or significant disease progression.

ELIGIBILITY:
Inclusion Criteria:

ARM A and B: Phase I CP-4055 single agent 1. Patients must have relapsed/refractory leukemias for which no standard therapies are anticipated to result in a durable response or have failed potentially curative therapy, or have refused or are considered unsuitable for standard therapy

ARM C: CP-4055 in combination with idarubicin

1. Patients with relapsed/refractory AML for which no standard therapies are anticipated to result in a durable response or who have failed potentially curative therapy, or who refuse or are considered unsuitable for standard therapy

   ARM A, B, C: CP-4055 as single agent and/or in combination with idarubicin
2. Patients must be 18 years of age or older
3. Patients must have ECOG performance status (PS) of 0 - 2. See Appendix 3
4. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must have a negative serum or urine pregnancy test within 2 weeks prior to beginning treatment on this study. Nursing patients are excluded.

   Male and female patients must use acceptable contraceptive methods for the duration of time on study, and males also for 3 months after the last CP-4055 dose
5. Patients must be capable of understanding and complying with parameters as outlined in the protocol, and able and willing to sign a written informed consent form
6. In the absence of rapidly progressing disease, the interval from prior treatment to time of study drug administration should be at least 2 weeks for cytotoxic agents, or at least 5 half-lives for noncytotoxic agents.
7. Patients must have the following clinical laboratory values:

   * Serum creatinine less or equal to 1.5 x the institutional upper limit of normal (ULN)
   * Total bilirubin less or equal to 1.5 x the ULN unless considered due to Gilbert's syndrome
   * Alanine aminotransferase (ALT) (SGPT), or aspartate aminotransferase (AST) (SGOT) less or equal to 2.5 x the ULN unless considered due to organ leukemic involvement

Phase II

1. Patients with a confirmed diagnosis of AML who have received cytotoxic chemotherapy

2 - 7. Identical to inclusion criteria nos. 2 - 7 for phase I

Exclusion Criteria:

Phase I AND II

1. A history of allergic reactions or sensitivity attributed to compounds of similar chemical or biologic composition to CP-4055, i.e., ara-C and/or egg
2. Known positive status for human immunodeficiency virus (HIV) or hepatitis B or C
3. Pregnant and nursing patients are excluded
4. Uncontrolled intercurrent illness
5. Active heart disease
6. Patients receiving any other standard or investigational cytotoxic treatment for their hematologic malignancy other than a maximum of 5 g of hydroxyurea to a maximum of 5 days in cycle 1 of therapy
7. Any medical condition which in the opinion of the investigator places the patient at an unacceptably high risk for toxicities

   Exclusion criteria no. 8 applies only in arm C:
8. Patients with hypersensitivity to idarubicin or any other component of the product, and/or other anthracyclines or anthracenediones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2006-05; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Phase I: Determine the MTD and PK properties of CP-4055 single agent. | Q4 2007
Phase II: Determine the efficacy of CP-4055 single agent in AML | Q4 2007

SECONDARY OUTCOMES:
Phase I: Evaluate the safety profile of CP-4055 single agent. | Q4 2007
Determine the MTD and PK of CP-4055 in combination with idarubicin. | Q2 2008
Phase II: Extended evaluation of the safety profile of CP-4055 single agent in AML | Q2 2008

CONTACTS AND LOCATIONS:
Overall Officials: Francis J Giles, MD, Principal Investigator — Institute for Drug Development (IDD), Cancer Therapy and Research Center, San Antonio, Texas, USA
Locations (16):
- United States (5):
  - Mew York Medical College, Division of Oncology, Valhalla, New York
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Institute for Drug Development (IDD), Cancer Therapy and Research Center, 7979 Wurzbach Rd., San Antonio, Texas
- France (4):
  - Hematology Service, Hôpital Beaujon and Hôpital Avicenne, Bobigny, Paris
  - Centre Hospitalier Universitaire, CHU de Lyon, Service d'Hematologie Clinique, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre Hospitalier Universitaire CHU de Toulouse, Hopital Purpan, Toulouse
- Germany (3):
  - University Hospital Benjamin Franklin Med.Clinic III, Berlin
  - Department of Internal Medicine Klinikum der Johann Wolfgang Goethe-Universität Medizinische Klinik II, Frankfurt am Main
  - Westfälische Wilhelms-Universität Münster Medizinische Klinik und Polikinik Innere Medizin A, Münster
- Italy (2):
  - Institute of Hematology & Medical Oncology L and A Serágnoli University of Bologna, Bologna
  - Universitá degli Studi di Roma Ematologia- Policlinico Tor Vergata, Rome
- Department of Hematology, Ullevål University Hospital, University of Oslo, Oslo, Norway
- Christie Hospital, Manchester, United Kingdom